CLINICAL TRIAL: NCT01588886
Title: Institute of Emergency and Critical Care Medicine , School of Yang-Ming University
Brief Title: Proton Pump Inhibitor Use is Associated With High Risk of Pneumonia in Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 101013-E
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2013-11

CONDITIONS: Chronic Kidney Disease; Pneumonia
Keywords: Proton pump inhibitors; Pneumonia; Retrospective cohort study
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with PPI: CKD with PPI use, follow up at least 5 years began PPI use
- with or without Pneumonia outcome: Patients were eligible for inclusion if they received any PPIs treatment between January 1, 1998 and December 31, 2002 and had been diagnosed with pneumonia between January 1, 1998 and December 31, 2008 in an inpatient setting.

SUMMARY:
Chronic kidney disease is a severe medical problem in Taiwan public health issue, which the highest incidence and prevalence rate in the world.Proton pump inhibitors may increase the risk of pneumonia appearance, which were caused by profound irreversible gastric acid suppression. The study purpose was to characterize difference of developing pneumonia in chronic kidney disease of prior use proton pump inhibitors.

DETAILED DESCRIPTION:
The study used data from Taiwan Health Insurance Research Database; the investigators conducted a population-based cohort study in Taiwan. Case consisted of all patients who had a first diagnosis of chronic kidney disease for the period between 1997 and 2008. The investigators utilized the use of Proton pump inhibitor from chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease

Exclusion Criteria:

* excluded those patients who had ever been diagnosed with CKD before 1997

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investiators use the longitudinal health insurance database 2008 (LHID 2008) released by the Taiwan National Health Research Institutes (NHRI) in 2009. Taiwan implemented its National Health Insurance (NHI) program in 1995 to provide affordable health care for all the island's residents.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Chronic kidney disease ICD-9 | 2012-Dec

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chih-Hung, MD, Study Director — west-garden Hospital

REFERENCES:
- [Result] Sheen E, Triadafilopoulos G. Adverse effects of long-term proton pump inhibitor therapy. Dig Dis Sci. 2011 Apr;56(4):931-50. doi: 10.1007/s10620-010-1560-3. Epub 2011 Mar 2. PMID 21365243
- [Result] Wu H, Jing Q, Wang J, Guo X. Pantoprazole for the prevention of gastrointestinal bleeding in high-risk patients with acute coronary syndromes. J Crit Care. 2011 Aug;26(4):434.e1-6. doi: 10.1016/j.jcrc.2010.12.007. Epub 2011 Jan 26. PMID 21273036
- [Result] Madanick RD. Proton pump inhibitor side effects and drug interactions: much ado about nothing? Cleve Clin J Med. 2011 Jan;78(1):39-49. doi: 10.3949/ccjm.77a.10087. PMID 21199906